CLINICAL TRIAL: NCT07097272
Title: Sternal Closure Techniques in High-BMI Patients Undergoing Open-Heart Surgery: A Retrospective Observational Comparison of Cable and Wire Systems
Brief Title: Sternal Closure in High-BMI Patients: Cable vs Wire
Status: Active, not recruiting | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SamsunKVC SCW
Record Dates: First submitted 2025-06-25; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-06

CONDITIONS: Sternal Wound Complications; Obesity (Body Mass Index >30 kg/m2); Median Sternotomy; Cardiac Surgery
Keywords: Cardiac Surgery; Postoperative Complications; Sternum Closure; Sternal Cable; Sternal Wire
MeSH Terms: conditions — Obesity; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard wire group: Patients with BMI ≥30 who underwent median sternotomy and had sternal closure using standard stainless-steel wire.
- cable system group: Patients with BMI ≥30 who underwent median sternotomy and had sternal closure using the RTI Surgical Sternal Cable System.

SUMMARY:
This retrospective study compares two sternal closure techniques-standard stainless-steel wires and rigid cable systems-in adult patients with a body mass index (BMI) ≥30 who underwent open-heart surgery between January 1, 2020, and December 31, 2024. The study aims to evaluate the incidence of sternal instability, wound infections, reoperation, and length of stay in the intensive care unit and hospital. Findings may help inform surgical decision-making for high-BMI patients.

DETAILED DESCRIPTION:
Elevated body-mass index (BMI ≥ 30 kg/m²) is an established risk factor for sternal wound complications after median sternotomy, yet consensus is lacking on the optimal closure technique in this high-risk subgroup. Conventional monofilament stainless-steel wiring remains the worldwide standard because it is inexpensive and familiar, but multifilament cable systems provide greater fatigue strength and more uniform load distribution in bench testing and early clinical reports. Previous meta-analyses report conflicting results-some indicating fewer sternal complications with rigid fixation, others showing no clear benefit-largely because they pool heterogeneous populations in which obesity is often only one of many overlapping risk factors. The present study isolates the effect of BMI by retrospectively analysing all adult patients (≥18 years) with BMI ≥ 30 kg/m² who underwent primary open-heart surgery at a single tertiary centre from 1 January 2020 through 31 December 2024. Patients are stratified by the sternal closure method actually used-standard simple/figure-of-eight wires versus a commercially available rigid cable system (RTI Surgical Sternal Cable). By excluding other indications for rigid fixation (eg, age ≥ 80, dialysis, osteoporosis, COPD, bilateral internal mammary harvest, mediastinitis, early re-exploration, re-do sternotomy), the analysis aims to discern whether obesity alone modifies the relative performance of the two techniques. De-identified peri-operative data are extracted from electronic records under institutional ethics approval, and pre-specified statistical comparisons will quantify associations between closure method and postoperative sternal instability, surgical site infection, need for reoperation, and resource utilisation (ICU and total hospital length of stay). Findings are expected to refine evidence-based recommendations for sternal closure in high-BMI cardiac-surgery patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Body Mass Index (BMI) ≥30 kg/m²
3. Underwent primary open-heart surgery via median sternotomy
4. Sternal closure performed with either standard stainless-steel wire or multifilament sternal cable system
5. Complete and accessible perioperative clinical records

Exclusion Criteria:

1. Age ≥80 years
2. End-stage renal disease or chronic hemodialysis
3. Redo sternotomy
4. Early postoperative re-exploration (within 7 days)
5. Mediastinitis prior to index discharge
6. Diabetic patients with bilateral internal mammary artery (IMA) harvest
7. Diagnosed osteoporosis
8. Chronic obstructive pulmonary disease (FEV₁ <80% and FEV₁/FVC <70%)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients (≥18 years) with a body mass index (BMI) of 30 kg/m² or higher who underwent primary open-heart surgery via median sternotomy at a single tertiary cardiovascular surgery center. All patients received sternal closure using either standard stainless-steel wire or a rigid multifilament cable system. Patients with additional indications for rigid sternal fixation-such as advanced age, dialysis, reoperation, or osteoporosis-were excluded to isolate the effect of BMI on outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Sternal Instability and Major Wound Complications | 90 days after surgery
  This outcome measures the rate of sternal instability (e.g., dehiscence, nonunion, displacement requiring intervention) and major sternal wound complications (e.g., deep sternal wound infection, mediastinitis, or reoperation for closure failure) in patients with BMI ≥30 undergoing open-heart surgery. The results will be compared between patients whose sternum was closed with standard stainless-steel wire versus those treated with a multifilament sternal cable system.

SECONDARY OUTCOMES:
Intensive Care Unit Length of Stay | Postoperative Day 0 through ICU discharge, up to 14 days
  Number of days from admission to discharge in the intensive care unit (ICU) following open-heart surgery.
Total Hospital Length of Stay | Postoperative Day 0 through hospital discharge, up to 30 days
  Total number of days from surgery to hospital discharge, reflecting overall resource utilization.
Reoperation Not Related to Sternal Closure Failure | 30 days postoperatively
  Incidence of any surgical re-intervention within 30 days postoperatively for causes unrelated to sternal instability (e.g., bleeding, tamponade).

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun University Faculty of medicine, Samsun, Turkey (Türkiye)